CLINICAL TRIAL: NCT01947543
Title: Calmodulin Gene Mutations in Patients With Ventricular Arrhythmia of Unknown Origin - A Screening Study
Status: Withdrawn | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Ole Frobert, MD, PhD, MD, PhD, Region Örebro County
Other Study IDs: Protocol no: 2012-11
Record Dates: First submitted 2013-08-27; First posted 2013-09-20 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ventricular tachycardia: Patients with ventricular tachycardia of unknown origin treated with an ICD.
- Family members: Family members (parents, siblings and children) for patients with results showing mutations in the calmodulin genes.

SUMMARY:
The aim of this study is to screen a well characterized patient population with ventricular tachycardia of unknown origin and treated with an implantable cardioverter-defibrillator (ICD) for mutations in the calmodulin genes.

DETAILED DESCRIPTION:
Patients with ventricular tachycardia of unknown origin and treated with an implantable cardioverter-defibrillator (ICD) will be asked to participate in the study. For patients with results showing mutations in the calmodulin genes, family members (parents, siblings and children) will also be asked to participate in the study. For under age patients and relatives who agree to participate, informed consent will also be taken from their custodian.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ventricular tachycardia of unknown origin that have been treated with an ICD
* Signed and dated informed consent

Exclusion Criteria:

- Inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ventricular tachycardia of unknown origin and treated with an ICD
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Mutations in the calmodulin genes | 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Fröbert, MD, Ph.D., Principal Investigator — Department of Cardiology, Örebro University Hospital, Örebro, Sweden
Locations (1):
- Department of Cardiology, Örebro University Hospital, Örebro, Sweden